CLINICAL TRIAL: NCT04463329
Title: Is Jedi Grip Efficient And Effective In Ultrasound Guided Peripheral Nerve Block: A Prospective, Randomized, Observer-Blinded Comparison Between Single And Double Operator Technique
Brief Title: Jedi Grip vs. Double Operator Technique for Axillary Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-18-1955
Record Dates: First submitted 2020-07-04; First posted 2020-07-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Brachial Plexus Block; Ultrasound, Interventional
Keywords: Brachial Plexus Block, Ultrasound-Guided, Jedi Grip, Double operator peripheric nerve block

STUDY DESIGN:
Intervention Model Description: the patients were randomly allocated to one of the two groups as Group C (conventional two-operator axillary brachial plexus blockage) and Group J (axillary brachial plexus block with single operator using Jedi grip)
Who Masked: Outcomes Assessor
Masking Description: After completion of the block, a blinded observer recorded demographic data and questioned the patients for felt pain related to the block procedure using a 10-cm visual analog scale (0 cm = no pain, 10 cm = worst imaginable pain). Patients were also questioned for symptoms related to the local anesthetic toxicity.
  Subsequently, measurements of brachial plexus blockade were carried out every 5 mins until 30 mins by the same blinded observer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): conventional two-operator axillary brachial plexus blockage
  Interventions: Procedure: conventional two-operator versus single operator using Jedi grip axillary brachial plexus blockage
- Group J (Active Comparator): axillary brachial plexus block with single operator using Jedi grip
  Interventions: Procedure: conventional two-operator versus single operator using Jedi grip axillary brachial plexus blockage

INTERVENTIONS:
Procedure: conventional two-operator versus single operator using Jedi grip axillary brachial plexus blockage — on goup C, operator used the probe and needle with different hands while an assistant controlling the syringe to aspirate or inject local anesthetic. On Group J single operator controlled the probe with one hand while controlling the needle and the syringe on the other hand with the Jedi technique. The needle was held between the index finger and the middle phalanx of the middle finger, and the syringe was held with fingers 4 and 5, with the plunger part to the thumb in the palm.

SUMMARY:
In this prospective randomized controlled observer-blinded study we aimed to compare the efficacy of a single operator technique so called Jedi Grip and conventional technique requiring double operator in ultrasound guided axillary brachial plexus block.

DETAILED DESCRIPTION:
Patients aged between 18 and 65 years, American Society of Anesthesiologists (ASA) physical status I to II ) undergoing elective hand, wrist and forearm surgery were prospectively enrolled. Patients were randomly assigned to Group C (conventional technique) or group J (Jedi technique). In both groups, axillary plexus blockage was provided by applying 5cc of a mixture of 10 cc 0.5% bupivacaine and 10 cc 2% prilocaine to the ulnar, radial, median and musculocutaneous nerves. Parameters such as performance time and the number of needle passes were recorded during procedure. Subsequently, a blinded observer evaluated and recorded parameters related to the success of blockage. The main outcome variable was performance time and success rate (surgical anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective hand, wrist and forearm surgery

Exclusion Criteria:

* hepatic or renal failure, serious cardiac or pulmoner disease, local or systemic infection, sepsis, coagulation disorder, neurological, muscular or psychiatric disease, body mass index (BMI) below 18.5 or above 35, drug and substance abuse, pregnancy, refusal of regional anesthesia, history of allergy to local anesthetics, mental-motor retardation (inability to consent or assess the visual analog scale(VAS) pain score), preoperative long-term NSAIDs or opioid use and prior surgery in the axillary regions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
block performance time | during procedure
  the sum of imaging and needling times
success rate | during operation
  patients percentage with provided successful anesthesia

SECONDARY OUTCOMES:
Onset time of sensory block | before operation
  Sensory blockage was evaluated and graded; from lateral to the forearm, the volar face of the thumb, volar face of the 5th finger and lateral side of the hand back; for musculocutaneous, median, ulnar and radial nerves, respectively. Graduation was according to 3-point scale using a cold test: 0 = no block, 1 = analgesia (patient can feel touch, not cold), and 2 = anesthesia (patient cannot feel touch).
Onset time of motor block | before operation
  Motor blockage was evaluated and graded; with elbow flexion, thumb abduction, thumb opposition, thumb adduction for musculocutaneous, radial, median, ulnar nerves respectively. Motor blockage graduation was also according to a 3-point scale: 0 = no block, 1 = paresis and 2 = paralysis.[

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Aytac, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pappin D, Christie I. The Jedi Grip: a novel technique for administering local anaesthetic in ultrasound-guided regional anaesthesia. Anaesthesia. 2011 Sep;66(9):845. doi: 10.1111/j.1365-2044.2011.06845.x. No abstract available. PMID 21831086